CLINICAL TRIAL: NCT02022540
Title: A Phase I Open-Label, Multi-Center Trial With Randomization to Dose to Evaluate the Safety and Tolerability of Topical Ocular PAN-90806 in Patients With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Phase 1 Study of Topical Ocular PAN-90806 for Neovascular AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PanOptica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAN-01-101
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Age-Related Macular Degeneration (AMD)
Keywords: Neovascular Age-Related Macular Degeneration; AMD; Macular Degeneration; Age-Related Macular Degeneration; wet AMD; neovascular AMD; exudative AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Stage 1 - Group 1 (Experimental): Patients randomized to Group 1 will receive PAN-90806 Ophthalmic Solution daily for 8 weeks.
  Interventions: Drug: PAN-90806 Ophthalmic Solution
- Stage 1 - Group 2 (Experimental): Patients randomized to Group 2 will receive PAN-90806 Ophthalmic Solution daily for 8 weeks.
  Interventions: Drug: PAN-90806 Ophthalmic Solution
- Stage 1- Group 3 (Experimental): Patients randomized to Group 3 will receive PAN-90806 Ophthalmic Solution daily for 8 weeks.
  Interventions: Drug: PAN-90806 Ophthalmic Solution
- Stage 1- Group 4 (Experimental): Patients randomized to Group 4 will receive PAN-90806 Ophthalmic Solution daily for 8 weeks.
  Interventions: Drug: PAN-90806 Ophthalmic Solution
- Stage 1 - Group 5 (Experimental): Patients randomized to Group 5 will receive PAN-90806 Ophthalmic Solution daily for 8 weeks.
  Interventions: Drug: PAN-90806 Ophthalmic Solution
- Stage 2 (Experimental): Patients enrolled in Stage 2 will receive an intravitreal injection of ranibizumab and then 7-9 days later begin daily dosing with PAN-90806 Ophthalmic Solution for 12 weeks
  Interventions: Drug: PAN-90806 Ophthalmic Solution; Drug: Lucentis

INTERVENTIONS:
Drug: PAN-90806 Ophthalmic Solution
  Other Names: PAN-90806 Eye Drops
Drug: Lucentis
  Other Names: ranibizumab
  Arms: Stage 2

SUMMARY:
The objective of this study is to assess the safety and tolerability of topical ocular PAN-90806 in patients with active, subfoveal choroidal neovascularization associated with neovascular Age-Related Macular Degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis in the study eye of active, pathologic, newly diagnosed and previously untreated, subfoveal choroidal neovascular (CNV) lesions secondary to neovascular AMD
* Aged 50 years or older
* Demonstrate the ability, or have a family member who is willing and able, to instill topical ocular drops in the study eye

Exclusion Criteria:

* No prior ocular or systemic treatment or surgery for neovascular AMD in the study eye
* History of or current clinical evidence in the study eye of:

  * aphakia
  * diabetic macular edema
  * any ocular inflammation or infections
  * pathological myopia
  * retinal detachment
  * advanced glaucoma
  * significant media opacity, including cataract
* History or evidence of the following surgeries in the study eye:

  * penetrating keratoplasty or vitrectomy;
  * corneal transplant;
  * corneal or intraocular surgery within 3 months of Screening
* Uncontrolled hypertension despite use of antihypertensive medications
* Participation in any investigational drug or device study, systemic or ocular, within past 3 months
* Women who are pregnant or nursing
* Known serious allergies or hypersensitivity to the fluorescein dye used in angiography or to the components of the PAN-90806 formulation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months
  Presence of any targeted adverse events (TAEs); safety endpoints include adverse events, vital signs, laboratory abnormalities, ophthalmic findings and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wax, M.D., Study Director — PanOptica, Inc.
Locations (22):
- United States (22):
  - Colorado Springs, Colorado
  - Winter Haven, Florida
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Boston, Massachusetts
  - Portsmouth, New Hampshire
  - Bloomfield, New Jersey
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Statesville, North Carolina
  - Ashland, Oregon
  - Philadelphia, Pennsylvania
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Harlingen, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Willow Park, Texas
  - Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided